CLINICAL TRIAL: NCT04915053
Title: Black Garlic Nutraceuticals Supplementation for the Control of Blood Pressure in Hypertension. A Triple-blind Randomized Placebo Control Study.
Brief Title: Black Garlic Nutraceuticals and Blood Pressure Control
Acronym: ENDOGARLIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat de Lleida (Other)
Collaborators: Pharmactive, S.L. (Unknown)
Responsible Party: Principal Investigator, José Serrano, Principal Investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIC-2435
Record Dates: First submitted 2021-05-24; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: Garlic; Nitric oxide; Angiotensin-converting enzyme; Antioxidant capacity; Endothelial function
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Three measurements, initial, middle, and final.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Random number of samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABG Black Garlic Extract (Experimental): Daily intake of a 550 mg tablet, containing 250 mg of Black Garlic Extract and 300 mg of excipients.
  Interventions: Dietary Supplement: ABG+ Black Garlin
- Placebo (Placebo Comparator): Daily intake of a 550 mg tablet, containing 250 mg of microcrystalline cellulose and 300 mg of excipients
  Interventions: Dietary Supplement: Crystalline Cellulose

INTERVENTIONS:
Dietary Supplement: ABG+ Black Garlin — Daily tablet intake during three months
  Arms: ABG Black Garlic Extract
Dietary Supplement: Crystalline Cellulose — Daily tablet intake during three months
  Arms: Placebo

SUMMARY:
Black garlic contains a series of allyl-sulfur compounds with the ability to modulate nitric oxide synthetase, angiotensin-converting enzyme system, and endothelial activation, which together could help better control blood pressure. The main objective of this study is to evaluate the effect on blood pressure and endothelial health of a daily intake of a black garlic supplement named ABG (registered mark), which has a higher concentration of black garlic bioactive compounds, in people with moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

- Clinical hypertension, medically treated with no more than 2 drugs

Exclusion Criteria:

* Body mass index above 35 kg/m2
* Fasting blood cholesterol levels below 115 mg/dL
* Fasting blood glucose levels above 126 mg/dL
* Taking anyone of the Angiotensin-converting enzyme inhibitors
* Anemia (hemoglobin below 13 g/dL in men and below 12 g/dL in women)
* Vitamin or nutraceutical intake in the last 30 days before the study enrollment
* Chronic gastrointestinal diseases
* Pregnancy and breastfeeding
* Garlic allergy
* Participation in another study 30 days before the study enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure | Baseline and 12 weeks
  Indirect measure of blood pressure by a trained physician

SECONDARY OUTCOMES:
Change in Blood nitric oxide content | Baseline and 12 weeks
  Nitric oxide determined by nitrate and nitrite content in blood
Change in Angiotensin-converting enzyme activity | Baseline and 12 weeks
  Activity measured by a substrate-enzyme activity kit
Change in Endothelial function | Baseline and 12 weeks
  Endothelial blood flow capacity
Change in Blood lipid profile | Baseline and 12 weeks
  Analysis of lipid profile (Total-cholesterol, LDL-cholesterol, Triacylglycerides, HDL-Cholesterol)
Change in Blood cytokine profile | Baseline and 12 weeks
  Analysis of cytokine profile (TNFa, IL-1b, IL-18, IL-6, IL-8, IL-17, IL-23, TGFb) in blood by immunoassays (Multiplexed)
Change in Blood antioxidant capacity | Baseline and 12 weeks
  Reduction capacity of blood determined by a biochemistry assay

CONTACTS AND LOCATIONS:
Overall Officials: Manuel S Portero, PhD, Principal Investigator — Universitat de Lleida
Locations (1):
- Hospital Arnau de Vilanova, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared.